CLINICAL TRIAL: NCT03090529
Title: The Role of Exercise Training in the Treatment of Resistant Hypertension
Acronym: EnRIcH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: University Institute of Maia (Other); Cardiology Department, Hospital Infante D. Pedro, Centro Hospitalar do Baixo Vouga (Unknown); Hypertension and Cardiovascular Unit, Hospital Pedro Hispano, ULS Matosinhos (Unknown); Cintesis & Departamento de Medicina da Faculdade de Medicina do Porto (Unknown)
Responsible Party: Principal Investigator, Fernando Ribeiro, Adjunct Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1725/2014
Record Dates: First submitted 2017-03-13; First posted 2017-03-24 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Resistant Hypertension
Keywords: Exercise training; Ambulatory blood pressure; Resistant Hypertension; Nitric Oxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The 12-week exercise-training program will include three sessions of aerobic exercise per week
  Interventions: Other: Exercise Group
- Control group (No Intervention): The control group will receive usual medical care

INTERVENTIONS:
Other: Exercise Group — The 12-week exercise-training program will include three sessions of aerobic exercise per week
  Arms: Exercise group

SUMMARY:
The main purpose of this study is to assess whether exercise training reduces ambulatory blood pressure in patients with resistant hypertension. To accomplish these goals 60 patients with resistant hypertension will be recruited and randomized into exercise training or control groups and followed up for 6 months. The patients in the exercise group will participate in a 3-month outpatient program. The control group will receive usual medical care. At baseline, after the intervention and 3 months after the end of the intervention both groups will undergo several evaluations, including casual and ambulatory blood pressure, body composition, cardiorespiratory fitness, quality of life, arterial stiffness, autonomic function, and endothelial and inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria: confirmed resistant hypertension, who in the previous 3 months had unchanged medication

Exclusion Criteria:

1. Patients with secondary hypertension
2. Evidence of target organ damage
3. Patients with heart failure
4. Previous cardiovascular event
5. Peripheral artery disease
6. Renal failure
7. Chronic obstructive pulmonary disease
8. Systolic office blood pressure superior to 180 mmHg
9. Biomechanical limitations to physical activity
10. Those participating in regular physical activity

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure | Change from Baseline in Blood Pressure at 3 months
  Blood pressure

SECONDARY OUTCOMES:
Casual blood pressure | Change from baseline to 3 months
  Blood pressure
Body composition | Change from baseline to 3 months
  Body composition
Health-related quality of life | Change from baseline to 3 months
  Health-related quality of life will be evaluated by the Short-Form 36.
Arterial stiffness | Change from baseline to 3 months
  Carotid-femoral pulse wave velocity, central pressures and aortic augmentation index and augmentation pressure.
Heart rate variability | Change from baseline to 3 months
  Recordings of R-R interval data; The R-R interval will be analyzed using time domain, frequency domain and Poincare´ plot techniques.
Circulating number of endothelial progenitor cells, circulating endothelial cells, nitric oxide and endothelial Nitric Oxide Synthase | Change from baseline to 3 months
  These markers will inform endothelial function, damage and repair
Inflammation | Change from baseline to 3 months
  Plasma levels of inflammatory and anti-inflammatory biomarkers.
Oxidative stress | Change from baseline to 3 months
  Plasma levels of oxidative stress and antioxidant markers.
Daily physical activity | Change from baseline to 3 months
  Physical activity will be measured during 7 consecutive days using an accelerometer.
Dietary intake | Change from baseline to 3 months
  Dietary intake will be assessed using a 4-day food diary.
VO2 max | Change from baseline to 3 months
  VO2 max will be determined by the Chester step test.

CONTACTS AND LOCATIONS:
Overall Officials: José Mesquita Bastos, MD, PhD, Study Director — Hospital Infante D. Pedro, Centro Hospitalar Do Baixo Vouga
Locations (2):
- Portugal (2):
  - Cardiology Department, Hospital Infante D. Pedro, Centro Hospitalar do Baixo Vouga, Aveiro
  - Hypertension and Cardiovascular Unit, Hospital Pedro Hispano, ULS Matosinhos, Matosinhos Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopes S, Mesquita-Bastos J, Garcia C, Bertoquini S, Ribau V, Teixeira M, Ribeiro IP, Melo JB, Oliveira J, Figueiredo D, Guimaraes GV, Pescatello LS, Polonia J, Alves AJ, Ribeiro F. Effect of Exercise Training on Ambulatory Blood Pressure Among Patients With Resistant Hypertension: A Randomized Clinical Trial. JAMA Cardiol. 2021 Nov 1;6(11):1317-1323. doi: 10.1001/jamacardio.2021.2735. PMID 34347008